CLINICAL TRIAL: NCT03193112
Title: Melatonin Decreases Eye Pressure in Depressive Patients With Normal Intraocular Pressure
Brief Title: Melatonin Decreases Eye Pressure in Normotensive Patients
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gokhan Ozdemir, Principal investigator, Clinical Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: KahramanmarasSIU
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Depressive Disorder
Keywords: Agomelatine; Depression; Intraocular pressure
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — agomelatine; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- Study group: The investigators analyze the intraocular pressure changes on patients who have been using Agomelatine for their primary depressive disorder. For the treatment of depression, patients will have been started routinely Agomelatine tablet of 25 mg orally. The investigators measure the eye pressure for one months in those patients receiving standard depression treatment.
  Interventions: Drug: Agomelatine 25 MG Oral Tablet

INTERVENTIONS:
Drug: Agomelatine 25 MG Oral Tablet — We will treat our patients with Agomelatine tablet of 25 mg.

SUMMARY:
Agomelatine is a melatonin drug used to treat depressive disorder. Agomelatine may also some effects on ocular pressures. In this study, we aimed to demonstrate that melatonin decreases intraocular pressures when given depressive patients.

DETAILED DESCRIPTION:
Melatonin has been shown to be effective to decrease intraocular pressure in experimental animal researches. Agomelatine is a melatonin derivative drug approved for the treatment of depression, which is also available in our country. Depending on animal experiments, it can be assumed that agomelatine can decrease intraocular pressure. Demonstrating that agomelatine is effective to reduce eye pressure may give a concurrent treatment of depressive patients with glaucoma. With this it may be possible to treat both diseases at the same time with single drug. In this study, the researchers intended to investigate the changes in ocular tension in normotensive depressive patients treated with agomelatine.

ELIGIBILITY:
Inclusion Criteria:

* Depressive patients suitable for Agomelatine therapy for the treatment of their primary disease.

Exclusion Criteria:

- Any past history of ocular surgery, ocular trauma or existing ocular diseases

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators seek to analyze the intraocular pressure changes depending on Agomelatin treatment. Depressive patients who are deemed suitable for agomelatine treatment on a routine basis by psychiatry clinic will be monitored with regard to intraocular pressure changes. Treatment decision will be given by the psychiatrist independently from patient's enrollment to the study. Then, investigators will measure intraocular pressure before the treatment and one month after the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | One month
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Ozdemir, MD, Principal Investigator — KSU
Locations (1):
- Kahramanmaras Sutcuimam University Ophthalmology Department, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No